CLINICAL TRIAL: NCT04699149
Title: Combining rTMS and Video Game-based Dexterity Training to Improve Dexterity in Parkinson's Disease: a Randomized Controlled Pilot-study
Brief Title: Combining rTMS and Video Game-based Dexterity Training to Improve Dexterity in Parkinson's Disease
Acronym: rTMSVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKNZ 2019-00433
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: transcranial magnetic stimulation; dexterity; video game-based training
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: blinded randomised clinical trial
Who Masked: Participant
Masking Description: rTMS protocol either sham or real
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): The PD patients randomized in the experimental group will receive VBT each time preceded by a real rTMS stimulation.
  Interventions: Other: Transcranial magnetic stimulation
- sham stimulation (Sham Comparator): The PD patients randomized in the control group will receive VBT each time preceded by a sham TMS.
  Interventions: Other: Sham transcranial magnetic stimulation

INTERVENTIONS:
Other: Transcranial magnetic stimulation — Non-invasive brain stimulation
  Arms: real stimulation
Other: Sham transcranial magnetic stimulation — Non-invasive brain stimulation
  Arms: sham stimulation

SUMMARY:
We investigate the effectiveness of a combined repetitive transcranial magnetic stimulation (rTMS) - video game-based training (VBT) dexterity intervention in Parkinson's diseases. The short and long-term benefits of this training program will be evaluated. For these purposes, a blinded sham controlled randomized controlled trial will be performed.

DETAILED DESCRIPTION:
Patients with Parkinson's disease (PD) often exhibit dexterous difficulties during the performance of activities of daily living (ADL) such as tying shoe laces, hand-writing, using remote controls, smartphone or tablet. These difficulties further add to the burden of the disease, leading to reduced quality of life (QoL). A relatively new, but rapidly growing aspect of training in PD neurorehabilitation is exergaming. To enhance training effects a combination of repetitive transcranial magnetic stimulation (rTMS) with exergaming will be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed PD
2. Hoehn & Yahr I to IV
3. Age 50-80 years old
4. written and signed informed consent
5. dexterous difficulties-

Exclusion Criteria:

1. Significant medical, psychiatric co-morbidity including dementia as defined by Montreal Cognitive Assessment (MOCA < 21)
2. Inability to understand the scope of the study and to follow study procedures according to the protocol e.g. complete questionnaires (i.e. due to cognitive problems)
3. Exclusion criteria for TMS and Sham application, such as current pregnancy, personal history of epilepsy or epileptic fits, and any psychiatric, neurologic, or medical history.
4. Participation in another interventional trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
DextQ-24 | 3 weeks
  standardized patient self-rated outcome measure (PROM) for evaluating dexterity related ADL in PD

SECONDARY OUTCOMES:
Nine Hole Peg test (9-HPT) | 3 weeks
  The 9-HPT is a standardized, well established, and reliable measure of hand dexterity in patients with PD.
Coin rotation task (CRT) | 3 weeks
  The CRT measures fine coordinated finger movements and is a suitable and valid dexterity test in patients with PD.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanbellingen, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pastore-Wapp M, Kaufmann BC, Nyffeler T, Wapp S, Bohlhalter S, Vanbellingen T. Feasibility of a combined intermittent theta-burst stimulation and video game-based dexterity training in Parkinson's disease. J Neuroeng Rehabil. 2023 Jan 12;20(1):2. doi: 10.1186/s12984-023-01123-w. PMID 36635679
- [Derived] Pastore-Wapp M, Lehnick D, Nef T, Bohlhalter S, Vanbellingen T. Combining Repetitive Transcranial Magnetic Stimulation and Video Game-Based Training to Improve Dexterity in Parkinson's Disease: Study Protocol of a Randomized Controlled Trial. Front Rehabil Sci. 2021 Nov 23;2:777981. doi: 10.3389/fresc.2021.777981. eCollection 2021. PMID 36188867